CLINICAL TRIAL: NCT00119431
Title: Pharmacokinetics, Clinical Efficacy and Safety of C1 Inhibitor Concentrate (C1-Esteraseremmer-N) for the Treatment of Hereditary (and Acquired) Angioedema
Brief Title: Kinetics, Efficacy and Safety of C1-Esteraseremmer-N
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KB2003.01A
Record Dates: First submitted 2005-07-04; First posted 2005-07-13 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Hereditary Angioedema Type I; Angioneurotic Edema
Keywords: Hereditary angioedema type I (MeSH: angioneurotic edema, complement 1 inactivators)
MeSH Terms: conditions — Hereditary Angioedema Types I and II; Angioedema

INTERVENTIONS:
Drug: C1 inhibitor concentrate

SUMMARY:
A multicentre study to investigate pharmacokinetics, clinical efficacy and safety of nanofiltered Cetor® (called C1-esteraseremmer-N during the development phase) for the treatment of hereditary angioedema (HAE) will be performed. This study KB2003.01 consists of three parts, part A pharmacokinetics (phase II), part B treatment of attacks of angioedema (phase III) and part C prophylactic use of C1 inhibitor (phase III). Part B + C will provide data on the efficacy of C1-esteraseremmer-N.

The changes in the manufacturing process of C1-esteraseremmer-N, compared to Cetor® (the currently marketed C1-inhibitor product), nanofiltration and omission of hepatitis B immunoglobulin, most likely will not affect tolerability. The nanofiltration will provide more safety regarding viruses.

In part A, the pharmacokinetics of C1-esteraseremmer-N in patients with hereditary angioedema will be compared with the current registered product, Cetor®, in a randomised, blinded cross-over design. This study has to provide evidence that changes in the manufacturing process have not affected pharmacokinetics. In addition, this study provides data on safety of C1-esteraseremmer-N.

DETAILED DESCRIPTION:
A multicentre study to investigate pharmacokinetics, clinical efficacy and safety of nanofiltered Cetor® (called C1-esteraseremmer-N during the development phase) for the treatment of hereditary angioedema (HAE) will be performed. This study KB2003.01 consists of three parts, part A pharmacokinetics (phase II), part B treatment of attacks of angioedema (phase III) and part C prophylactic use of C1 inhibitor (phase III). Part B + C will provide data on the efficacy of C1-esteraseremmer-N.

The changes in the manufacturing process of C1-esteraseremmer-N, compared to Cetor® (the currently marketed C1-inhibitor product), nanofiltration and omission of hepatitis B immunoglobulin, most likely will not affect tolerability. The nanofiltration will provide more safety regarding viruses.

In part A, the pharmacokinetics of C1-esteraseremmer-N in patients with hereditary angioedema will be compared with the current registered product, Cetor®, in a randomised, blinded cross-over design. This study has to provide evidence that changes in the manufacturing process have not affected pharmacokinetics. In addition, this study provides data on safety of C1-esteraseremmer-N. Twelve HAE patients without signs of an attack will receive an administration of 1,000 U, 1,500 U or 2,000 U of C1-esteraseremmer-N or Cetor® and later on the same dose of the other product. Both antigenic and functional C1 inhibitor levels will be determined. Laboratory safety parameters and adverse events will be monitored as well

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of hereditary angioedema type I: i.e. markedly decreased C1 inhibitor activity, decreased level of C1 inhibitor antigen and a decreased level of C4.
* Age ≥ 18 years
* Body weight between 40 and 100 kg.
* Signed Informed consent

Exclusion Criteria:

* C1 inhibitor infusion within the last 7 days
* Signs of any attack
* Angioedema attack within 7 days before actual infusion of study medication
* Change in the dosage of androgens in the last 14 days before the study
* Change in oral anticonceptive medication in the last two months before the study
* Pregnancy or lactation.
* B-cell malignancy
* Participation in another pharmaceutical clinical study, which can interfere with this study, in the last 3 months prior to the study
* History of clinically relevant antibody development to C1 inhibitor
* Use of oral anticoagulant medication in the last 14 days
* Use of heparin within the last two days prior to the study
* History of allergic reaction to C1 inhibitor concentrate or other blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of C1-esteraseremmer-N versus Cetor.

SECONDARY OUTCOMES:
Laboratory and clinical safety as well as clinical tolerance of C1-esteraseremmer-N versus current Cetor.

CONTACTS AND LOCATIONS:
Overall Officials: M. M. Levi, Prof. Dr., Principal Investigator — Academic Medical Centre Amsterdam
Locations (2):
- Netherlands (2):
  - Academic Medical Centre, Amsterdam
  - Erasmus Medical Centre, Rotterdam